CLINICAL TRIAL: NCT00038649
Title: Therapy of Early Chronic Phase Chronic Myelogenous Leukemia (CML) With Higher-Dose Gleevec (STI571)
Brief Title: Therapy of Early Chronic Phase CML With Higher-Dose Gleevec, Alpha Interferon, and Low-Dose Ara-C
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor discontinued providing study drug.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID01-151
Record Dates: First submitted 2002-06-03; First posted 2002-06-04 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-09

CONDITIONS: Myelogenous Leukemia, Chronic, Chronic Phase
Keywords: Philadelphia chromosome positive; early chronic phase (diagnosis < 12 months); Chronic Myelogenous Leukemia, Chronic Phase; Chronic Myelogenous Leukemia; CML; Gleevec; STI571
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gleevec (Experimental): Gleevec 400 mg orally twice daily.
  Interventions: Drug: Gleevec

INTERVENTIONS:
Drug: Gleevec — 400 mg orally twice daily
  Other Names: imatinib mesylate; STI-571

SUMMARY:
The goal of this clinical research study is to see if higher doses of imatinib mesylate (Gleevec, STI571) can improve chronic myelogenous leukemia (CML) in chronic phase.

DETAILED DESCRIPTION:
Imatinib mesylate is a new oral medication that blocks a protein that is responsible for CML

Before treatment starts, patients will have a physical exam, blood tests, and a bone marrow study. The bone marrow will be removed with a large needle. Women able to have children will have a screening blood or urine test for pregnancy.

Patients on this study will take 400 mg of imatinib twice daily (morning and evening). If you have side effects, the dose may be lowered. If you are taking less than 800 mg of imatinib, you can take your dose once per day or divided in two doses. Imatinib mesylate should be taken with a large glass of water. Bottles containing the tablets will be given to the patient every 6 months. Unused supplies must be returned at the end of the study.

After completing 3 to 12 months of therapy, response to imatinib mesylate will be evaluated. If the response is good, treatment with imatinib mesylate alone will be continued. Treatment may be continued for up to 20 years, or as long as it is judged best to control the leukemia.

Update: June 2010 Blood tests are recommended 2 times per year. Your doctor will discuss with you how often you should have blood tests. Bone marrow will be done if your doctor thinks it is necessary to check your disease. You must return to MD Anderson at least once every year. You may not need a bone marrow test every visit, but you will have blood drawn to measure the amount of disease you have. If the leukemia cannot be found for 2 years or longer on the blood test called polymerase chain reaction (PCR) which is done to measure the amount of disease you have, your doctor may talk to you about stopping treatment with imatinib. If you and your doctor decide to stop your therapy, you will have a blood test for PCR done every 3 to 6 months. You do not need to return to MD Anderson to have this blood test done. You may have the blood taken by your local doctor and mailed to M. D. Anderson. If the leukemia is found again by the PCR blood test, your doctor may recommend that you restart treatment with imatinib. You may decide to stay on treatment with imatinib even if your PCR blood test does not show any sign of leukemia for 2 years or longer.

This is an investigational study. Imatinib mesylate has been approved in CML. A total of 125 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age 15 years or older with a diagnosis of Ph-positive or Bcr-positive CML in early chronic phase CML (diagnosis < 12 months). Except for hydroxyurea, patients must have received no or minimal prior therapy, defined as less than 1 month of prior interferon (IFN-a) or ara-C.
2. Eastern Cooperative Oncology Group (ECOG) performance of 0-2
3. Serum bilirubin less than 2 mg%, serum creatinine less than 2mg%
4. Women of pregnancy potential must practice contraception. Women and men must continue birth control for the duration of the trial and at least 3 months after the last dose of study drug.
5. Patients must sign an informed consent indicating they are aware of the investigational nature of this study, in keeping with the policies of the hospital.
6. The definitions of CML phases are as follows: a) early chronic phase: time from diagnosis to therapy < 12 months, late chronic phase: time from diagnosis to therapy > 12 months; b) blastic phase: presence of 30% blasts or more in the peripheral blood or bone marrow; c) accelerated phase CML: presence of any of the following features: peripheral or marrow blasts 15% or more, peripheral or marrow basophils 20% or more, thrombocytopenia <100 x 10(9)/L unrelated to therapy, documented extramedullary blastic disease outside liver or spleen due to past causes
7. The definitions of CML phases are as follows: clonal evolution defined as the presence of additional chromosomal abnormalities other than the Ph chromosome is part of accelerated phase CML. Ph chromosome variants or complex Ph chromosome translocations are not considered to indicate disease acceleration. We have recently found clonal evolution to have a variable prognostic impact and may be suppressed with IFN-a therapy. Hence these patients will be eligible if no other accelerated phase signs are present, and analyzed separately.
8. Inclusion of women and minorities: As per NIH policy, women and members of minorities will be included in this protocol as they are referred in the CML population. Their distribution is similar to the general referral profiles for CML: about 50% of CML patients are females and 25% to 30% are members of minorities. There are no exclusions of women or minorities based on the study objectives.

Exclusion Criteria:

1. New York Heart Association (NYHA) class 3-4 heart disease
2. Psychiatric disability (psychosis)
3. Pregnant or lactating females
4. Patients in late chronic phase, accelerated phase or blastic phase are excluded.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2001-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Cortes, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Jain P, Kantarjian H, Boddu PC, Nogueras-Gonzalez GM, Verstovsek S, Garcia-Manero G, Borthakur G, Sasaki K, Kadia TM, Sam P, Ahaneku H, O'Brien S, Estrov Z, Ravandi F, Jabbour E, Cortes JE. Analysis of cardiovascular and arteriothrombotic adverse events in chronic-phase CML patients after frontline TKIs. Blood Adv. 2019 Mar 26;3(6):851-861. doi: 10.1182/bloodadvances.2018025874. PMID 30885996
- [Derived] Issa GC, Kantarjian HM, Gonzalez GN, Borthakur G, Tang G, Wierda W, Sasaki K, Short NJ, Ravandi F, Kadia T, Patel K, Luthra R, Ferrajoli A, Garcia-Manero G, Rios MB, Dellasala S, Jabbour E, Cortes JE. Clonal chromosomal abnormalities appearing in Philadelphia chromosome-negative metaphases during CML treatment. Blood. 2017 Nov 9;130(19):2084-2091. doi: 10.1182/blood-2017-07-792143. Epub 2017 Aug 23. PMID 28835440
- [Derived] Jain P, Kantarjian H, Nazha A, O'Brien S, Jabbour E, Romo CG, Pierce S, Cardenas-Turanzas M, Verstovsek S, Borthakur G, Ravandi F, Quintas-Cardama A, Cortes J. Early responses predict better outcomes in patients with newly diagnosed chronic myeloid leukemia: results with four tyrosine kinase inhibitor modalities. Blood. 2013 Jun 13;121(24):4867-74. doi: 10.1182/blood-2013-03-490128. Epub 2013 Apr 25. PMID 23620574
- See also: University of Texas MD Anderson Cancer Center Official Website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: June 11, 2001 to April 25, 2003. All recruitment done in medical settings at University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the 117 participants enrolled, three were excluded before starting: two (2) withdrew from the study prior to initiation of treatment and one (1) was ineligible.
Period: Overall Study
Arm/Group | Gleevec
Started | 114
Completed | 105
Not Completed | 9
Not completed — Adverse Event | 9

BASELINE CHARACTERISTICS:
Arm/Group | Gleevec
Number analyzed (Participants) | 114
Age, Continuous [Median (Full Range); unit: years] | 48 [17 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 71
Region of Enrollment [Number; unit: participants]
  United States | 114

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Molecular Response of Complete or Partial Hematologic Remission
Description: Complete Hematologic Remission (CHR): normalization >4 weeks of bone marrow (<5% blasts), peripheral blood with White Blood Cells (WBC) <10 x 109/L & no peripheral blasts, promyelocytes or myelocytes; disappearance all signs/symptoms disease. Partial Hematologic Response (PHR) = CHR except persistence of immature cells (myelocytes, metamyelocytes), or splenomegaly < 50% of pretreatment, or thrombocytosis >450x109/L but <50% of pretreatment. Hematologic surveys twice per year with bone aspirations at discretion of treating physician.
Time Frame: Response to imatinib mesylate evaluated after completing 3 - 12 months of therapy.
Measure: Number; unit: participants
Arm/Group | Gleevec
Number analyzed (Participants) | 114
participants
  CHR | 110
  PHR | 0

2. Secondary Outcome: Participant Complete Hematologic Remission (CHR) Classified
Description: Number of participants with Complete Hematologic Remission (CHR): normalization >4 weeks of bone marrow (<5% blasts), peripheral blood with WBC <10 x 109/L & no peripheral blasts, promyelocytes or myelocytes; disappearance all signs/symptoms disease. CHR further classified according to suppression of Philadelphia chromosome (Ph) by cytogenetics or i Fluorescence In Situ Hybridization (FISH): No cytogenetic response - Ph positive 100% of pretreatment value; Minor cytogenetic response - Ph positive 35-90% of pretreatment value; Partial cytogenetic response - Ph positive 1-34% of pretreatment value; Complete cytogenetic response - Ph positive 0%. Hematologic surveys twice per year with bone aspirations at discretion of treating physician.
Time Frame: Response to imatinib mesylate evaluated after completing 3 - 12 months of therapy.
Population: Analysis was of the 110 participants who achieved a CHR with a cytogenetic response as described in the outcome measure descriptions.
Measure: Number; unit: participants
Arm/Group | Gleevec
Number analyzed (Participants) | 110
participants
  No cytogenetic response | 0
  Minor cytogenetic response | 1
  Partial cytogenetic response | 4
  Complete cytogenetic response | 105

ADVERSE EVENTS:
Time Frame: Total duration of therapy anticipated to be 15-20 years. Adverse events were collected from initiation of treatment, every 6 months yearly. Overall study period was June 2001 to August 2013.
Arm/Group | Gleevec
Serious Adverse Events (participants affected / at risk) | 45/114
Other Adverse Events (participants affected / at risk) | 59/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gleevec (N=114)
Death (General disorders) | 4 (4)
Arthritis (Cardiac disorders) | 1 (1)
Bleeding (Blood and lymphatic system disorders) | 1 (1)
Cardiac Arrythmia (Cardiac disorders) | 1 (1)
Cardiac; NOS (Cardiac disorders) | 1 (1)
Cardiovascular Accident (Cardiac disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Diarrhea/Vomiting (Gastrointestinal disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Eye Irritation (Eye disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1)
Hip Replacement Surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
Increased Liver Enzymes (Hepatobiliary disorders) | 1 (1)
Left Ventricular Systolic Dysfunction (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Prolapse Colon (Gastrointestinal disorders) | 1 (1)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rotator cuff Repair (Surgical and medical procedures) | 1 (1)
Ruptured Ovarian Cyst (Reproductive system and breast disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Small Bowel Obstruction (Gastrointestinal disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Surgery (Surgical and medical procedures) | 1 (1)
Surgery Abdominal Mass (Surgical and medical procedures) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Gallbladder disorder - Cholecystectomy (Gastrointestinal disorders) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 2 (2)
Fever (Investigations) | 2 (2)
Left Ventricular Diastolic Dysfunction (Cardiac disorders) | 1 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pregnancy (Reproductive system and breast disorders) | 2 (2)
Atrial Fibrallation (Cardiac disorders) | 3 (3)
Depression (Nervous system disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Gastroenteritis (Gastrointestinal disorders) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Elective Surgery (Surgical and medical procedures) | 5 (6)
Pain (General disorders) | 7 (7)
Secondary Malignancy (General disorders) | 7 (8)
Infection (Infections and infestations) | 9 (10)
Angioplasty (Cardiac disorders) | 1 (1)
Coronary artery bypass grafting (CABG) required (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gleevec (N=114)
Chest Pain (Cardiac disorders) | 9 (9)
Vomiting (Gastrointestinal disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Infection (Infections and infestations) | 9 (10)
Elective Surgery (Surgical and medical procedures) | 6 (7)
Pain (General disorders) | 7 (7)
Secondary Malignancy (General disorders) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes